CLINICAL TRIAL: NCT06581419
Title: A Phase I/II Clinical Study Evaluating Safety, Tolerability, and Efficacy of IAP0971 in Advanced Tumors
Brief Title: A Clinical Trial to Evaluate Effect of IAP0971 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IAP0971-203
Record Dates: First submitted 2024-08-22; First posted 2024-09-03 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Advanced Malignant Neoplasm; Advanced or Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phase I (Experimental): Dose escalation (Phase I): 14 to 48 subjects with advanced malignancies are planned to be enrolled to initially investigate the safety and tolerability of IAP0971 and to determine the MTD based on the frequency of DLT in each dose arm.The starting dose of IAP0971 for injection is 0.0005 mg/kg, with a preset maximum escalation dose of 18.0 mg/kg, administered once every 3 weeks.
  Interventions: Drug: IAP0971
- phase II (Experimental): Dose Extension (Phase II) : Phase II will use an open-label, non-randomized, single-arm, multicenter design. Under the RP2D dose determined in Phase I, 20-30 untreated patients with advanced or metastatic non-small cell lung cancer, who are driver gene negative and PD-L1 positive (TPS ≥ 50%), will be enrolled. The drug IAP0971 is administered once every 3 weeks, and every 3 weeks is 1 cycle
  Interventions: Drug: IAP0971

INTERVENTIONS:
Drug: IAP0971 — Subjects receive IAP0971, which will be administered every 3 weeks in a 3-week cycle.

SUMMARY:
Phase I: To evaluate the safety, tolerance and effectiveness of IAP0971 for the treatment of advanced malignant tumors.

Phase II: Evaluation of IAP0971 therapy driver negative and PD-L1 positive (TPS≥50%) The initial treatment is effective in subjects with advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
The study includes dose-escalation (Phase I) and dose-expansion (Phase II) clinical trials. Phase I clinical trials will be conducted first. After completing the dose-escalation phase, the plan is to determine the recommended Phase II dose (RP2D) in the maximum tolerated dose (MTD) group and proceed with the subsequent Phase II exploratory studies.

The objective of the Phase I dose-escalation phase is to preliminarily assess the safety and tolerability of IAP0971 and to determine the MTD based on the incidence of dose-limiting toxicities (DLTs) in each dose group. Phase II will use an open-label, non-randomized, single-arm, multicenter design. The study will evaluate adverse events and adverse reactions through clinical observation, vital sign monitoring, and laboratory tests. Tumor assessments will be conducted using RECIST 1.1 criteria: within 48 weeks of the first infusion of the investigational drug, assessments will be performed after every two cycles (±7 days), and after 48 weeks, assessments will occur every four cycles (±7 days) until disease progression, initiation of new anti-tumor therapy, investigator-determined ineligibility (e.g., intolerable adverse reactions), loss to follow-up, voluntary withdrawal, death, or study termination/suspension.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years old (including cut-off value), regardless of gender.
2. Phase I only: patients with histologically confirmed advanced or metastatic malignant solid tumors who have failed to respond to standard treatment, who have no standard treatment options, who are not currently applicable to standard treatment, or who have been assessed by the investigator to benefit from this treatment.
3. Phase II only: patients with histologically confirmed locally advanced (stage IIIB or IIIC) or metastatic (stage IV) non-small cell lung cancer (NSCLC) that is not amenable to complete surgical resection and definitive concurrent chemoradiotherapy. Note: For patients with locally advanced stage (stage IIIB/IIIC) who cannot accept radical concurrent/sequential chemoradiotherapy, they need to be evaluated by relevant professional physicians and confirmed by written records.
4. Phase II only: no prior systemic antitumor therapy for locally advanced or metastatic NSCLC (except for patients who received adjuvant/neoadjuvant chemotherapy or definitive concurrent or sequential chemoradiotherapy for locally advanced disease and disease progression ≥6 months after the last treatment).
5. Phase II only: PD-L1 positive (TPS≥50%) as determined by IHC, and patients were negative for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) by immunohistochemistry.
6. have at least one measurable lesion according to RECIST 1.1 criteria (tumor lesion located in the previous radiotherapy area or other locoregional treatment site, generally not considered a measurable lesion unless the lesion has clearly progressed or persists beyond three months of radiotherapy).
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
8. predicted survival time ≥3 months.
9. with adequate organ function:

   ① Blood system (no blood transfusion or hematopoietic stimulation therapy within 14 days) : absolute neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥100×109/L, hemoglobin (HGB) ≥90 g/L; ② Liver function: total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN), except Gilbert's syndrome Out of; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 times ULN, and patients with liver metastasis or liver cancer need AST and ALT≤5.0 times ULN and total bilirubin ≤3.0 times ULN;

   ② Renal function: serum creatinine (Cr) ≤1.5 times ULN; If creatinine > 1.5 times ULN, creatinine clearance (Ccr) ≥50 mL/min (calculated by Cockcroft-Gault formula) was required.

   ③ Coagulation function: prothrombin international normalized ratio (INR) ≤1.5 times ULN, activated partial thromboplastin time (APTT) ≤1.5 times ULN, patients with liver metastasis or liver cancer need INR and APTT≤2.5 times ULN.
10. Eligible patients (men and women) of childbearing potential must consent to use a reliable method of contraception (hormonal or barrier methods or abstinence) with their partner during the trial and for at least 6 months after the last dose; Female patients of reproductive age had to have a negative blood pregnancy test within 7 days before the first use of the study drug.
11. Subjects must give informed consent for this study and voluntarily provide written informed consent before the trial.

Exclusion Criteria:

1. Phase II only: small cell lung cancer or sarcomatoid lesion confirmed by histopathology.
2. Phase II only: previous immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1 /PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonists (e.g. ICOS, CD40, CD137, GITR, OX40 antibody, etc.), immune cell therapy, and any treatment targeting the mechanism of tumor immune action.
3. Phase I only: patients received anti-tumor therapy such as systemic chemotherapy, radiotherapy, biological therapy, endocrine therapy, or immunotherapy within 4 weeks before the first dose of study drug; The following drugs were excluded according to the following criteria:

   ① Treatment with a small-molecule tyrosine kinase inhibitor within 2 weeks before the first dose;

   ② Palliative local treatment for non-target lesions within 2 weeks before the first dose; Patients received non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, not including IL-11) within 2 weeks before the first dose;

   ③ received Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 2 weeks before the first dose.
4. received other investigational drugs or treatments within 4 weeks before the study drug.
5. received systemic glucocorticoids (prednisone > 10 mg/ day or equivalent) or other immunosuppressive agents within 14 days before the first dose of study drug; The use of topical, ocular, intra-articular, nasal, and inhaled glucocorticoids was excluded. Short-term prophylaxis with glucocorticoids (e.g., to prevent contrast allergy).
6. the adverse effects of previous antineoplastic therapy have not recovered to CTCAE 5.0 grade ≤1 or the relevant requirements of the inclusion criteria (except for toxicities without safety risks judged by the investigators, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stable with hormone replacement therapy).
7. major surgical procedures (excluding needle biopsies) within 4 weeks before the first dose of study drug, major trauma, or the need for elective surgery during the trial.
8. prior allogeneic hematopoietic stem-cell transplantation or organ transplantation.
9. clinically symptomatic parenchymal or meningeal metastases.
10. have active infection and currently require intravenous anti-infective therapy.
11. have a history of immunodeficiency, including testing positive for human immunodeficiency virus (HIV) antibodies.
12. active hepatitis B (HBsAg positive and HBV-DNA positive or greater than the upper limit of normal), active hepatitis C (hepatitis C virus antibody positive and HCV RNA positive or greater than the upper limit of normal).
13. received any live vaccine within 4 weeks before the first dose of study drug.
14. known hypersensitivity to any antibody-based drug (NCI CTCAE grade 5.0 ≥3) or to the study drug, active ingredient, or inactive excipients of a PD-1/PD-L1 inhibitor.
15. with severe and uncontrollable lung diseases (severe infectious pneumonia, interstitial lung disease, etc.); Or other moderate-to-severe lung diseases that severely affect respiratory function that may interfere with the detection or management of drug-related pulmonary toxicity.
16. have a history of severe cardiovascular and cerebrovascular disease, including but not limited to:

    ① Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular block, etc.

    ② Mean QT interval corrected with Fridericia's method (QTcF) > 470 ms;

    ③ Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months before the first dose; ④ patients with New York Heart Association (NYHA) functional class ≥II heart failure or left ventricular ejection fraction (LVEF) < 50% or structural heart disease with high risk as judged by other investigators; And 5) clinically uncontrolled hypertension.
17. have an active or previous autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) with the possibility of recurrence, except clinically stable autoimmune thyroid disease, type I diabetes mellitus, vitiligo, cured atopic dermatitis in children, and psoriasis (within the past 2 years) that does not require systemic treatment."
18. had other malignancies within 5 years before study administration, except for malignancies that could be expected to be cured with treatment (including, but not limited to, adequately treated thyroid cancer, carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with radical surgery).
19. have clinically uncontrollable effusion in the third space, which was judged by the investigator to be not suitable for enrollment.
20. known alcohol or drug dependence.
21. with mental disorders or poor adherence.
22. pregnant or lactating women.
23. The participant was deemed by the investigator to have a history of other serious systemic diseases or to be ineligible for the study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAEs (Phase I) | 3 months after end event visit
  To investigate the safety characteristics.progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data.
Dose limiting toxicities (DLTs) (Phase I) | 21 days after first dose
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D).
PFS in dose expansion (Phase II) | Baseline through up to 2 years or until disease progression
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1.

SECONDARY OUTCOMES:
pharmacokinetic parameters Cmax (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  Cmax after single administration
pharmacokinetic parameters Tmax (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  Tmax after single administration
pharmacokinetic parameters AUC 0-t (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  AUC 0-t after single administration
pharmacokinetic parameters AUC 0-∞ (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  AUC 0-∞ after single administration
pharmacokinetic parameters CL (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  CL after single administration
pharmacokinetic parameters Vd (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  Vd after single administration
pharmacokinetic parameters t1/2 (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  t1/2 after single administration
pharmacokinetic parameters λz (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  λz after single administration
pharmacokinetic parameters Css,max (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  Css,max after multiple administration
pharmacokinetic parameters Css,min (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  Css,min after multiple administration
pharmacokinetic parameters Css,av (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  Css,av after multiple administration
pharmacokinetic parameters AUCss (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  AUCss after multiple administration
pharmacokinetic parameters CLss (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  CLss after multiple administration
pharmacokinetic parameters Vss (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  Vss after multiple administration
pharmacokinetic parameters R (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  R after multiple administration
pharmacokinetic parameters DF (Phase I) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  DF after multiple administration.
Immunogenicity (Phase I) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAP0971.(Phase I)
Objective response rate (ORR) in dose escalation (Phase I) | Baseline through up to 2 years or until disease progression
  Tumor response based on RECIST 1.1.
ORR (Phase II) | Baseline through up to 2 years or until disease progression
  ORR as assessed using RECIST 1.1.
OS (Phase II) | Baseline through up to 2 years or until disease progression
  OS as assessed using RECIST 1.1.
DCR (Phase II) | Baseline through up to 2 years or until disease progression
  DCR as assessed using RECIST 1.1.
Incidence of AEs and SAEs (Phase II) | 3 months after end event visit
  To investigate the safety characteristics.
Incidence of ADA (Phase II) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAP0971

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No